CLINICAL TRIAL: NCT05338034
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group Phase 2a Study to Evaluate the Efficacy and Safety of HPG1860 in Subjects With Nonalcoholic Steatohepatitis
Brief Title: Phase 2a Study of HPG1860 in Subjects With NASH
Acronym: RISE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hepagene (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPG1860-201
Record Dates: First submitted 2021-10-24; First posted 2022-04-20 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During this study, subjects, investigators, the Sponsor, and the clinical research organization (CRO) (except specific vendors whose role in study conduct requires their unblinding, eg, personnel operationally associated with the interactive response technology [IRT]) will be blinded to the study intervention assignment. Study team personnel will remain blinded throughout the study with the exception of a Sponsor Committee who will review interim analysis results and make decisions regarding dropping and/or adding a treatment cohort and an unblinded study team member assigned to monitor that at least 6 subjects in each dose cohort had serial PK measurements taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HPG1860 3 mg (Experimental): 20 subjects will be treated with HPG1860 3 mg once daily at a similar time with or without food.
  Interventions: Drug: HPG1860
- HPG1860 5 mg (Experimental): 20 subjects will be treated with HPG1860 5 mg once daily at a similar time with or without food.
  Interventions: Drug: HPG1860
- HPG1860 8 mg (Experimental): 20 subjects will be treated with HPG1860 5 mg once daily at a similar time with or without food.
  Interventions: Drug: HPG1860
- Placebo (Placebo Comparator): 20 subjects will be treated with Placebo once daily at a similar time with or without food.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HPG1860 — The dosage form for clinical research is a dry-filled capsule for oral administration manufactured as strengths of 3 mg, 5 mg, and 8 mg.
  Arms: HPG1860 3 mg; HPG1860 5 mg; HPG1860 8 mg
Drug: Placebo — Capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2a, randomized, double-blind, placebo-controlled, parallel group, multiple arm, multicenter study of 3 different doses of HPG1860 versus placebo in subjects with biopsy-confirmed or phenotypic NASH.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled, parallel group, multiple arm, multicenter study of 3 different doses of HPG1860 versus placebo in subjects with biopsy-confirmed or phenotypic NASH. Screening will occur up to 5 weeks prior to randomization; all eligible subjects will have baseline hepatic imaging during Screening, prior to randomization. Approximately 80 eligible subjects will be randomized 1:1:1:1 on Day 1/Week 0 (T1) to receive either HPG1860 3 mg (n = 20), or 5 mg (n = 20), or 8 mg (n = 20), or placebo (n = 20) for 12 weeks. Following a preplanned interim analysis, a dose cohort may be dropped and/or added.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study-specific procedure.
2. Males and females between 18 and 75 years of age
3. Nonpregnant, nonlactating women.
4. Male subjects must agree to utilize a highly effective method of contraception.
5. Body mass index (BMI) of ≥25 kg/m2 at Screening.
6. Non-cirrhotic NASH subjects.
7. NASH subjects with hepatic fat assessed by a central reader
8. Willing and able to adhere to study restrictions and agree to comply with study protocol.

Exclusion Criteria:

1. Pregnant or lactating females
2. Current significant alcohol consumption
3. Elevated LDL-C with stable dose of statin an or PCSK9 inhibitor
4. Renal dysfunction or nephritic syndrome or a history of nephritis
5. Recent infarction, unstable angina leading to hospitalization, uncontrolled, symptomatic cardiac arrhythmia
6. Uncontrolled hypertension
7. Type 1 diabetes or uncontrolled T2DM
8. Uncontrolled hypothyroidism
9. Liver transplant and/or other significant liver disease or dysfunction
10. HIV antibody positive
11. Known hypersensitivity or formulation excipient
12. Gastrointestinal conditions or procedures that may affect drug absorption
13. Hematologic or coagulation disorders
14. Unstable weight within the last 3 months
15. Active malignancy
16. Unexplained creatine kinase (CK) >3 × ULN
17. Blood donation, blood transfusion
18. Unable to undergo or contraindication to MRI procedure
19. A medical or situational finding that in the investigator's opinion may compromise the subject's safety or ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males and females between 18 and 75 years of age; inclusive based on the date of Screening
Enrollment: 89 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of treatment | 12 weeks
  Number of participants Treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
liver fat content | 12 week
  Change from baseline (CFB) in liver fat content (LFC) measured by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) at Week 12
Percentage of subjects with ≥30% reduction in LFC from baseline | 4 week and 12 week
  measured by MRI-PDFF at Week 4 and Week 12
Change from baseline (CFB) in liver fat content (LFC) at 4 week | 4 week
  measured by MRI-PDFF at Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Naim Alkhouri, Principal Investigator — Arizona Liver Health - Tucson
Locations (1):
- South Texas Research Institute (STRI), Texas City, Texas, United States

IPD SHARING:
Plan to Share IPD: No
still pending